CLINICAL TRIAL: NCT04836546
Title: A Post Approval Study to Evaluate the Safety and Effectiveness of the Eversense® Continuous Glucose Monitoring (CGM) System Used Non-adjunctively
Brief Title: Eversense® Non-adjunctive Use Post Approval Study
Acronym: NA-PAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTP-0039
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Diabetes
Keywords: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Self monitoring of blood glucose, then CGM System (Experimental): All participants will first manage their diabetes with SMBG for 6 months followed by managing their diabetes with Eversense CGM system for the next 6 months
  Interventions: Device: Blood glucose meter; Device: Eversense CGM System

INTERVENTIONS:
Device: Blood glucose meter — First phase: SMBG for 6 months
Device: Eversense CGM System — Second phase: CGM for 6 months

SUMMARY:
This is a non-blinded, prospective, multi-center, single arm longitudinal cohort study (patient serving as their own control), to evaluate the effectiveness of diabetes with the Eversense CGM System non-adjunctively compared to self-monitoring of blood glucose (SMBG) using a blood glucose (BG) meter in participants with either Type 1 or Type 2 diabetes. Subjects will serve as their own control, with their baseline based on using SMBG to manage their diabetes for the first 6 months followed by using Eversense CGM System non-adjunctively for the second 6 months. Total follow-up duration is 12 months. The investigation will include both clinic visits and home use of Eversense CGM System. The nonadjunctive phase will have two sensors, up to 90-day duration, inserted sequentially. All care decisions specific to diabetes will be based on blood glucose (BG) values in the first phase and the Eversense CGM system values in the second phase.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has diabetes
2. Subject is ≥18 years of age
3. Subject has a smartphone that is internet enabled
4. Subject is able to comply with study protocol tasks and understand written and verbal instructions in the investigator's opinion
5. Subjects is willing and able to provide written signed and dated informed consent

Exclusion Criteria:

1. Subject is critically ill or hospitalized
2. Prior use of CGM defined as:

   * No more than 1 week of continuous CGM use in the last 6 months, and
   * At least 4 weeks of continuous use of CGM in the last 12 months or 12 weeks total use in the past 3 years.
3. Subject has a known contraindication to dexamethasone or dexamethasone acetate
4. Subjects requiring intravenous mannitol or mannitol irrigation solutions
5. Subject is on dialysis at the time of enrollment
6. Female subjects who are pregnant, planning on becoming pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 925 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate and severe hypoglycemic and diabetic ketoacidosis events | First 6 months (phase 1) compared to second 6 months (phase 2)
  Incidence of moderate and severe hypoglycemic and diabetic ketoacidosis events with SMBG use for 6 months compared to Eversense CGM system used non-adjunctively for 6 months

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - LA Universal Research Center, Inc., Los Angeles, California
  - Denver Endocrinology, Diabetes & Thyroid Center, Englewood, Colorado
  - CMR of Greater New Haven, Hamden, Connecticut
  - Chase Medical Research, Waterbury, Connecticut
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - MedCare Research, Miami, Florida
  - Miami Lakes Clinical Trials INC, Miami Lakes, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Springfield Clinic, Springfield, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - Southern Maryland Medical Group, Camp Springs, Maryland
  - Metro Detroit Endocrinology, Dearborn, Michigan
  - Diabetes and Endocinology Specialists, Inc., Chesterfield, Missouri
  - Endocrine Associates of West Village, Long Island City, New York
  - Physician's East Endocrinology, Greenville, North Carolina
  - Superior Clinical Research, Smithfield, North Carolina
  - AM Diabetes & Endocrinology, Bartlett, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Clinical Research Solution Institute, Houston, Texas
  - RGV Endocrine Center, McAllen, Texas
  - Green Mountain Research Institute, Rutland, Vermont

IPD SHARING:
Plan to Share IPD: No